CLINICAL TRIAL: NCT07316959
Title: Efficacy Of Long-Term Low Dose Macrolide Therapy In Preventing Early Recurrence Of Nasal Polyps After Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260/proposal-ENT/ERC
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps
Keywords: macrolides; Chronic Rhinosinusitis
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Received Macrolide (clarithromycin 250 mg) once day in addition to their usual prescription
  Interventions: Procedure: clarithromycin 250 mg
- Group B (Active Comparator): Patients in Group B received only their routine prescribed postoperative medications following surgery (no macrolide therapy).
  Interventions: Procedure: clarithromycin 250 mg

INTERVENTIONS:
Procedure: clarithromycin 250 mg — Following surgery, patients were split into two groups at random . For three months, patients in group A received Macrolide (clarithromycin 250 mg) once day in addition to their usual prescription drugs.
  Other Names: group B

SUMMARY:
This randomized controlled trial evaluated the effectiveness of long-term, low-dose clarithromycin (250 mg/day) in reducing symptoms, improving endoscopic and radiologic scores, and preventing early recurrence of nasal polyps after endoscopic sinus surgery. Conducted at the ENT Department of Sir Ganga Ram Hospital, Lahore, the study included patients aged 15-75 undergoing surgery for nasal polyps. Group A received clarithromycin for three months in addition to standard therapy, while Group B received standard therapy alone. Patients treated with clarithromycin showed significantly greater improvements in SNOT, Lund-Kennedy, and Lund-Mackay scores at 8 and 12 weeks compared to controls (p<0.05). Polyp recurrence at three months was also lower in the macrolide group (12%) than in the non-macrolide group (32%).

Overall, low-dose clarithromycin was found to be safe and effective in enhancing postoperative outcomes and reducing early recurrence of nasal polyps after endoscopic sinus surgery.

ELIGIBILITY:
Inclusion Criteria

Male and female patients aged 15 to 75 years

Clinical diagnosis of nasal polyps

Underwent endoscopic sinus surgery

Willing and able to provide informed consent Exclusion Criteria

Current or recent use of antibiotics or macrolide therapy

History of multiple facial fractures

Presence of neurological disorders

Presence of psychiatric or psychological disorders

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Change in symptom and disease severity scores | 3 months
  (Change in Sinonasal Outcome Test-22 (SNOT-22) , Lund-Kennedy score, and Lund-Mackay score) from baseline to 12 weeks after endoscopic sinus surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhammad Shouzib Sultan, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yamada T, Fujieda S, Mori S, Yamamoto H, Saito H. Macrolide treatment decreased the size of nasal polyps and IL-8 levels in nasal lavage. Am J Rhinol. 2000 May-Jun;14(3):143-8. doi: 10.2500/105065800782102717. PMID 10887619
- See also: Related Info — https://pesquisa.bvsalud.org/portal/resource/pt/wpr-172313